CLINICAL TRIAL: NCT02790021
Title: Improving the Quality of Life of Patients With Breast Cancer-related Lymphedema by Lymphaticovenous Anastomosis (LVA): A Randomized Controlled Trial
Brief Title: Microsurgical Treatment of Breast Cancer-related Lymphedema by Lymphaticovenous Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL67059.068.18
Record Dates: First submitted 2016-05-11; First posted 2016-06-03 (Estimated); Last update posted 2025-05-19 (Actual); Status verified 2025-05

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Complex decongestive therapy (No Intervention): Group A will continue complex decongestive therapy consisting of skin care, manual lymphatic drainage, and compression therapy using compression stockings.
- Lymphaticovenous anastomosis (LVA) (Experimental): Group B will undergo an LVA procedure under local anesthesia in surgical daycare setting. Patients are not allowed to wear compression stockings or have decongestive therapy for four weeks after the surgery.
  Interventions: Procedure: Lymphaticovenous anastomosis (LVA)

INTERVENTIONS:
Procedure: Lymphaticovenous anastomosis (LVA) — LVA is a minimally invasive procedure that can be performed under local anesthesia. Indocyanine green (ICG) lymphography is used to visualize the (obstructed) lymphatic vessels. When using the images as a guide, the lymphatic pathways and the sites for incisions for lymphaticovenous anastomoses are marked with a pen. The patient's limb is then prepared for surgery. Under a surgical microscope the lymphatic vessels are identified and viable lymphatic vessels are anastomosed to similarly sized adjacent recipient venules in the subdermal plane.
  Other Names: LVA
  Arms: Lymphaticovenous anastomosis (LVA)

SUMMARY:
Research question: Is lymphaticovenous anastomosis (LVA) for the treatment of breast cancer-related lymphedema of the arm (BCRL) more effective and cost-effective compared to standard conservative treatment? Hypothesis: LVA improves the health-related quality of life of patients who developed BCRL after breast cancer treatment and is cost-effective compared to conservative treatment. Study design: A multicenter randomised controlled trial (RCT) consisting of two treatment groups: conservative treatment (group A) and LVA (group B). The study is conducted in Maastricht University Medical Center, Radboud University Medical Center, Zuyderland Medical Center and Canisius-Wilhelmina Hospital. Study population: Women over 18 years old who underwent (axillary) treatment for breast cancer presenting with early stage lymphedema of the arm for which they received at least three months conservative treatment Intervention: LVA involves anastomosing lymphatic vessels to small veins to bypass obstructions in the lymphatic system.

Usual care: Complex decongestive therapy (CDT) which includes skin care, manual lymphatic drainage, and compression therapy. Outcome measures: The primary outcome is health-related quality of life after 12 months follow-up measured with the Lymph-ICF questionnaire. Secondary outcomes are (in)direct costs, QALYs, cost-effectiveness ratio, the discontinuation rate of conservative treatment, and excess limb volume. Sample size: A total of 120 patients will be included and randomised in two groups of 60 patients each.

Cost-effectiveness analysis: A trial-based economic evaluation is performed from the societal perspective to determine the cost-effectiveness, expressed in an incremental cost-effectiveness ratio (ICER) (i.e. cost per QALY gained), of LVA compared to CDT. Direct and indirect cost data is collected on the patient-level. The difference in QALYs is assessed with the EQ-5D-5L questionnaire. A Budget Impact Analysis (BIA) will be performed to analyse the financial consequences related to implementing LVA. Time schedule: Patient inclusion will take maximally 21 months. With a follow-up of 24 months, the total study period will be 48 months. The last three months are used for data analysis. Outcome assessment is at inclusion (before randomisation) and 3, 6, 12, 18, and 24 months later.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Treated for early stage breast cancer and who underwent an sentinel lymph node biopsy (SLNB), axillary lymph node dissection (ALND) or axillary radiotherapy
* Early stage lymphedema of the arm (ISL classification stage I/IIa; pitting edema without fibrosis) with viable lymphatic vessels as determined by indocyanin green (ICG) lymphography
* Already received at least three months of complex decongestive therapy (CDT) prior to inclusion
* Primary breast cancer
* Unilateral lymphedema
* Informed consent

Exclusion Criteria:

* Male sex
* Late stage lymphedema of the arm (ISL classification IIb/III lymphedema) with evident fat deposition and/or fibrosis
* History of earlier lymph reconstruction efforts
* Recurrent breast cancer
* Distant breast cancer metastases
* Bilateral lymphedema
* Primary congenital lymphedema
* Non-viable lymphatic system as determined by ICG lymphography

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life: Lymph-ICF questionnaire | 12 months
  To assess the efficacy of the treatment on disease-related symptoms we will use the "Lymphedema Functioning, Disability and Health" (Lymph-ICF)" questionnaire. This disease-specific questionnaire assesses the impairments in function, activity limitations, and participation restrictions of patients with arm lymphedema. This is a validated questionnaire, based on 5 domains with 29 questions. Each of the 29 questions corresponds to a score between 0-100. The total score on the Lymph-ICF is equal to the sum of the scores on the questions divided by the total number of answered questions. A higher score on the Lymph-ICF indicates more problems with functioning related to arm lymphedema.

SECONDARY OUTCOMES:
Cost-effectiveness of LVA compared to complex decongestive therapy | 24 months
  A trial-based economic evaluation is performed to determine the cost-effectiveness of LVA compared to complex decongestive therapy from the societal perspective. Cost data is collected on the patient-level and includes health care related costs, costs to patient and family, and costs due to lost productivity. The primary outcome measure for the effects is the quality-adjusted life year (QALY). Cost-effectiveness is expressed in an incremental cost-effectiveness ratio (ICER) (i.e. cost per QALY gained). In addition, a Budget Impact Analysis (BIA) will be performed from a budget holder perspective.
Excess limb volume | 24 months
  The relative arm volume is measured using the water displacement method (Bravometer), 3D volumetry, and circumference measurement. The volume of the affected arm is compared to the volume of the unaffected arm.
Discontinuation rate conservative therapy | 24 months
  The number of patients who are able to discontinue conservative therapy, i.e. no longer have to wear compression stockings or no more visits to the therapist, will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: René Van der Hulst, MD, PhD, Study Director — Maastricht University Medical Center; Shan Shan Qiu Shao, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Yasmine Jonis, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jonis YMJ, Wolfs JAGN, Hummelink S, Tielemans HJP, Keuter XHA, van Kuijk S, Ulrich DJO, van der Hulst RRWJ, Qiu SS. The 6 month interim analysis of a randomized controlled trial assessing the quality of life in patients with breast cancer related lymphedema undergoing lymphaticovenous anastomosis vs. conservative therapy. Sci Rep. 2024 Jan 26;14(1):2238. doi: 10.1038/s41598-024-52489-3. PMID 38278856
- [Derived] Wolfs J, Beugels J, Kimman M, Piatkowski de Grzymala AA, Heuts E, Keuter X, Tielemans H, Ulrich D, van der Hulst R, Qiu SS. Improving the quality of life of patients with breast cancer-related lymphoedema by lymphaticovenous anastomosis (LVA): study protocol of a multicentre randomised controlled trial. BMJ Open. 2020 Jan 15;10(1):e035337. doi: 10.1136/bmjopen-2019-035337. PMID 31948992